CLINICAL TRIAL: NCT06264635
Title: Pilot Randomized Controlled Trial Evaluating the Efficacy of Platelet-Rich-Plasma (PRP) for Erectile Dysfunction
Brief Title: Evaluating the Efficacy of Platelet-Rich-Plasma (PRP) for Erectile Dysfunction
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Premal Patel, MD, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS26227
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The provider and patient are both blinded to which treatment (PRP vs saline) the patient is receiving
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet-Rich-Plasma (PRP) (Experimental): PRP refers to a treatment where a patient's own blood is used to promote healing. Blood is drawn, processed to concentrate the platelets, and then re-injected into the injured area to stimulate tissue repair.
  Interventions: Biological: Platelet-Rich-Plasma
- Saline (Placebo Comparator): Provider will go through the same motions as injecting PRP, but will use saline instead which has no known effect.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Platelet-Rich-Plasma — PRP refers to a treatment where a patient's own blood is used to promote healing. Blood is drawn, processed to concentrate the platelets, and then re-injected into the injured area to stimulate tissue repair.
  Arms: Platelet-Rich-Plasma (PRP)
Other: Saline — Provider will go through the same motions as injecting PRP, but will use saline instead which has no known effect.
  Arms: Saline

SUMMARY:
There is great interest in restorative therapies (platelet-rich plasma (PRP) injections, shockwave therapy and stem cell therapy) for ED given their non-invasive nature. However, data is still limited and requires further research prior to widespread adoption. Unfortunately, therapies such as PRP injections are being widely used without clinical evidence demonstrating its safety or effectiveness for the treatment of erectile dysfunction. 2-7 To date, there are no treatments that address the underlying cause of endothelial dysfunction, although low-intensity shockwave therapy for ED has shown promising results. Platelet-derived therapies targeting inflammation and promoting tissue/nerve regeneration and may represent a potential treatment option towards this direction. The investigators propose to perform Canada's first pilot RCT to evaluate and safety and efficacy of PRP for the treatment of ED.

DETAILED DESCRIPTION:
The proposed study is a prospective, double-blinded, randomized placebo-controlled trial. This study will take place at the Manitoba Men's Health Clinic (Winnipeg, MB, Canada). All patients will undergo blood sampling in a 60 ml syringe containing 8 mL of anticoagulant. Patients will receive 2 treatments 1 month apart. Preparation of PRP and placebo injections will occur in a separate room. Samples of patients in the placebo arm will be discarded and sample of those randomized to the PRP group will be processed via an FDA-approved platelet separator (Magellan Autologous Platelet Separator; Arteriocyte Medical Systems, Hopkinton, MA) to yield approximately 10 mL of PRP. Once prepared, the patient will be placed in the supine position with a tourniquet placed around the base of the penis. A total of 5 mL will be infused in each corpus cavernosum - slowly retracting the needle for better distribution of PRP into the erectile tissue - over a 2-minute period. The whole procedure will be performed under sterile conditions. Following administration, additional compression of the penis will be performed with a dressing placed around the penile shaft. The penile tourniquet will be removed 20 minutes after the injections and patients are released. The placebo group will include a sterile saline injection. Follow-Up Procedures and Evaluations: Follow-up visits will be conducted at months: 1, 3, 6, after the last treatment session and shall include: Measuring IIEF-EF of patients at the clinic at every follow-up visit, as well as reporting and recording adverse events.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able willing and able to provide informed consent. The investigators wil enroll males between >30 and <70 years of age who have ED based on IIEF scores (score between 16 and 25.) with patients suffering from erectile dysfunction lasting for over 6 months and not more than 5 years as per history provided by patient.

The patient has been in a stable relationship for over 3 months prior to enrollment with a minimum of 2 sexual attempts per month for at least one month prior to enrollment.

A1C level ≤ 7% within 1 month prior to enrollment.

Exclusion Criteria:

* Participating in another study within the past three months that may interfere with the results or conclusions of this study, under judicial protection (prison or custody), adult under guardianship, or patient refuses to sign the consent.

History of radical prostatectomy or extensive pelvic surgery, past radiation therapy of the pelvic region within 12 months prior to enrolment, recovering from any cancer within 12 months prior to enrollment.

Neurological disease such as Alzheimer's or Parkinson's disease which affects erectile function at the discretion of the investigator, psychiatric diagnosis or medications such as antidepressants, anxiolytic, antipsychotic that affects erectile function or any other medications at the discretion of the investigator.

Anatomical malformation of the penis, including Peyronie's disease.

A1C level > 7% within 1 month prior to enrollment or history of Insulin dependent diabetes.

The patient is taking blood thinners and has an international normalized ratio (INR) >3.

Received shockwave treatment at least 6 months before enrollment.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) | 1, 3, 6 months post-procedure
  Follow-up visits will be conducted at months: 1, 3, 6, after the last treatment session and shall include: Measuring IIEF-EF of patients at the clinic at every follow-up visit. This is a validated form of assessing erectile function.

SECONDARY OUTCOMES:
Adverse Events | 1, 3, 6 months post-procedure
  Measuring and recording any adverse events post procedure such as hematomas, fibrosis, infections or worsening symptoms of erectile function.

CONTACTS AND LOCATIONS:
Locations (1):
- Men's Health Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No